CLINICAL TRIAL: NCT04779320
Title: A Randomized, Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of Vedolizumab Intravenous as Maintenance Therapy in Pediatric Subjects With Moderately to Severely Active Crohn's Disease Who Achieved Clinical Response Following Open-Label Vedolizumab Intravenous Therapy
Brief Title: A Study of Vedolizumab in Children and Teenagers With Moderate to Severe Crohn's Disease (CD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002-3025; 2020-004301-31 (EudraCT Number); jRCT2071210031 (Registry Identifier: jRCT); 2023-509045-13-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Crohn's Disease (CD)
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Induction Period: 10 to 15 kg, Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, intravenous (IV) infusion, at Day 1, Weeks 2 and 6 in Induction Period. Participants with CD having Baseline weight of 10 to 15 kg will be included in this arm group.
  Interventions: Drug: Vedolizumab IV
- Induction Period: >15 to <30 kg, Vedolizumab 200 mg (Experimental): Vedolizumab 200 mg, IV infusion, at Day 1, Weeks 2 and 6 in Induction Period. Participants with CD having Baseline weight of >15 to <30 kg will be included in this arm group.
  Interventions: Drug: Vedolizumab IV
- Induction Period: ≥30 kg, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, at Day 1, Weeks 2 and 6 in Induction Period. Participants with CD having Baseline weight of ≥30 kg will be included in this arm group.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: 10 to 15 kg Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, IV infusion, once every 8 weeks (Q8W) from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of 10 to 15 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 150 mg.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: 10 to 15 kg Vedolizumab 100 mg (Experimental): Vedolizumab 100 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of 10 to 15 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 100 mg.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: >15 to <30 kg, Vedolizumab 200 mg (Experimental): Vedolizumab 200 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of >15 to <30 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 200 mg.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: >15 to <30 kg Vedolizumab 100 mg (Experimental): Vedolizumab 100 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of >15 to <30 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 100 mg.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: ≥30 kg, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of ≥30 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 300 mg.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: ≥30 kg: Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of ≥30 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 150 mg.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV
  Other Names: ENTYVIO; KYNTELES; MLN0002

SUMMARY:
Vedolizumab is a medicine that helps to reduce inflammation and pain in the digestive system. In this study, children and teenagers with moderate to severe Crohn's disease will be treated with vedolizumab.

The main aim of the study is to check if participants achieve remission after treatment with the vedolizumab. Remission means symptoms improve or disappear and an endoscopy shows no signs of inflammation.

Participants will receive 3 infusions of vedolizumab over 6 weeks. Then, those who have a clinical response will receive either a high dose or low dose of vedolizumab once every 8 weeks. They will receive the same dose every time.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat pediatric participants who have moderately to severely active CD. The drug is tested and approved in adults in approximately 70 countries. Participants to be enrolled must have failed response to, lost response to, or been intolerant to at least 1 of the current standard of care (SOC) induction and maintenance therapies for CD including exclusive and/or partial enteral nutrition therapy, immunomodulators (e.g., azathioprine [AZA], 6-mercaptopurine [6-MP], methotrexate [MTX]), and tumor necrosis factor-alpha (TNF-α) antagonists.

The study will enroll approximately 120 patients.

During the Induction Period participants will receive 3 doses of vedolizumab IV infusion at Day 1, Week 2, and Week 6 based on their weight at Baseline as:

* Participants 10 to 15 kg, Vedolizumab 150 mg
* Participants >15 to <30 kg, Vedolizumab 200 mg
* Participants ≥30 kg, Vedolizumab 300 mg

At Week 14, participants who achieve clinical response will be randomly assigned (by chance, like flipping a coin) in a 1:1 ratio to one of the 2 double-blind dose groups (high dose and low dose), stratified by previous exposure/failure to TNF-α antagonists therapy or naive to TNF-α antagonists therapy, and by weight groups. Participants will receive vedolizumab IV infusions every 8 weeks (Q8W) up to Week 46 during the Maintenance Period as follows:

* Participants ≥30 kg, Vedolizumab 300 mg (High dose) or 150 mg (Low dose)
* Participants >15 to <30 kg, Vedolizumab 200 mg (High dose) 100 mg (Low dose)
* Participants 10 to 15 kg, Vedolizumab 150 mg (High dose) or 100 mg (Low dose)

The dose will remain blinded to the participant and study doctor during the study (unless there is an urgent medical need). All participants will be administered vedolizumab via IV infusion. In participants who demonstrate lack of maintenance of clinical response during the Maintenance Period the dose will be escalated in a blinded fashion to the high dose in their weight group based on the weight at the time of the worsening of disease. In addition one-time rescue therapy with corticosteroids is allowed during Maintenance Period.

This multi-center trial will be conducted worldwide. After the Week 54, participants may be eligible to continue receiving vedolizumab in extension study MLN0002-3029. Participants who do not maintain corticosteroid-free clinical response at week 54 will undergo an end-of-study (EOS) or ET visit, and a safety visit 18 weeks after the last dose of vedolizumab followed by 2 years of long term follow-up (up to 104 weeks), in addition these participants will then be eligible to enter study MLN0002-3029 for an observational LTFU period of 2 years after the last dose of study drug.

ELIGIBILITY:
Main Inclusion Criteria:

1. The participants has moderately to severely active CD, unresponsive or intolerant to their current standard of care (SOC).
2. The participants weigh ≥10 kg at the time of screening and enrollment into the study.
3. Participants with Crohn's disease (CD) diagnosed at least 1 month before screening. Participants with moderately to severely active CD defined by a Pediatric Crohn's Disease Activity Index (PCDAI) >30 and an simple endoscopic score for Crohn's Disease (SES-CD) >6 (or an SES-CD ≥4 if disease is confined to terminal ileum) at screening endoscopy.
4. Participants who have failed, lost response to, or been intolerant to treatment with at least 1 of the following agents: corticosteroids, immunomodulators (eg, azathioprine (AZA), 6-mercaptopurine (6-MP), methotrexate [MTX]), and/or tumor necrosis factor (TNF)-α antagonist therapy (eg, infliximab, adalimumab). This includes participants who are dependent on corticosteroids or exclusive or partial enteral nutrition to control symptoms and who are experiencing worsening of disease in the moderate-to-severe range when attempting to wean off corticosteroids or discontinue exclusive enteral nutrition.
5. Participants with extensive colitis or pancolitis of >8 years' duration or left-sided colitis of >12 years' duration must have documented evidence of a negative surveillance colonoscopy within 12 months before screening.
6. Participants with vaccinations that are up-to-date based on the countrywide accepted schedule of childhood vaccines.

Main Exclusion Criteria:

1. Participants who have received either (1) an investigational biologic (other than those listed in Exclusion Criterion #1) within 60 days or 5 half-lives before screening (whichever is longer); or (2) an approved biologic or biosimilar agent within 2 weeks before the first dose of study drug or at any time during the screening period.
2. Participants with active cerebral/meningeal disease, signs/symptoms or history of progressive multifocal leukoencephalopathy (PML) or any other major neurological disorders including stroke, multiple sclerosis, brain tumor or neurodegenerative disease.
3. The participants had a clinically significant infection (eg, pneumonia, pyelonephritis, coronavirus disease 2019 [COVID-19]) within 30 days prior to first dose of study drug.
4. The participants has received any live vaccinations within 30 days prior to first dose.
5. Participants who currently require surgical intervention or are anticipated to require surgical intervention for CD during this study.
6. Participants who have had subtotal or total colectomy or have a jejunostomy, ileostomy, colostomy, ileo-anal pouch, known fixed stenosis of the intestine, short bowel syndrome, or >3 small intestine resections.
7. Participants with a current diagnosis of indeterminate colitis.
8. Participants with clinical features suggesting monogenic very early-onset inflammatory bowel disease.
9. Active or latent tuberculosis (TB), as evidenced by a diagnostic TB test performed within 30 days of screening or during the screening Period that is positive, defined as:

   * Positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR
   * A TB skin test reaction ≥5 mm.
10. Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Hepatitis B virus (HBV) immune participants(i.e., hepatitis B surface antigen [HBsAg]-negative and hepatitis B antibody-positive) may, however, be included.

    Note: If a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if the absence of HBV DNA is confirmed by HBV DNA polymerase chain reaction reflex testing performed in the central laboratory.
11. Participants with chronic hepatitis C virus (HCV) (ie, positive HCV antibody [HCVAb] and HCV RNA).

    Note: Participants who are HCVAb-positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before baseline]).
12. The participants has any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
13. The participant has evidence of dysplasia or history of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
14. Participants with positive stool studies for ova and/or parasites or stool culture at screening visit.
15. Participants with positive Clostridioides difficile (C difficile) stool test at screening visit.

Other inclusion/exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Remission at Week 54 Based on Pediatric Crohn's Disease Activity Index (PCDAI) Score ≤10 | Week 54
  Clinical remission is defined by PCDAI score ≤10. The PCDAI was specifically designed for use in children. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: hematocrit (HCT) (adjusted for age and sex), erythrocyte sedimentation rate (ESR), and albumin level. The PCDAI score ranges from 0 to 100, with higher scores indicating more active disease. A score of <10 will be consistent with inactive disease, 11 to 30 will indicate mild disease, and >30 will indicate moderate to severe disease. A decrease of 12.5 points is taken as evidence of improvement.
Percentage of Participants With Endoscopic Response at Week 54 Based on Simple Endoscopic Score for Crohn's Disease [SES-CD] Score | Week 54
  Endoscopic response is defined as at least a 50% reduction in SES-CD score from Baseline. The overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables (ie, size of ulcers [cm], ulcerated surface, affected surface [%], and presence of narrowing) across 5 bowel segments (ie, rectum, descending and sigmoid colon, transverse colon, ascending colon, and ileum). Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is the most severe case, with the sum of the scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The segmental SES-CD score is the sum of the 4 variables for each bowel segment and can range from 0 to 12, where each individual variable score ranges from 0 to 3.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical and Endoscopic Remission at Week 14 Based on Both PCDAI Score and SES-CD Score | Week 14
  Clinical and endoscopic remission is where participant achieves both clinical and endoscopic remission. Clinical remission is defined by PCDAI score ≤10. Endoscopic remission is defined by SES-CD score of ≤4 with at least a 2-point reduction from Baseline and no sub-score >1. PCDAI includes child-specific item: height velocity variable as well as three laboratory parameters: HCT, ESR, albumin level. PCDAI score ranges from 0 to 100, with higher scores indicating more active disease. The SES-CD score ranges from 0 to 56 and is the sum of 4 variables, size of ulcers [cm], ulcerated surface, affected surface [%], and presence of narrowing) across 5 bowel segments (ie, rectum, descending and sigmoid colon, transverse colon, ascending colon, and ileum), where higher scores indicate more severe disease.
Percentage of Participants with Clinical and Endoscopic Remission at Week 54 Based on Both PCDAI Score and SES-CD Score | Week 54
  Clinical and endoscopic remission is where participant achieves both clinical and endoscopic remission. Clinical remission is defined by PCDAI score ≤10. Endoscopic remission is defined by SES-CD score of ≤4 with at least a 2-point reduction from Baseline and no sub-score >1. PCDAI includes child-specific item: height velocity variable as well as three laboratory parameters: HCT, ESR, albumin level. PCDAI score ranges from 0 to 100, with higher scores indicating more active disease. The SES-CD score ranges from 0 to 56 and is the sum of 4 variables, size of ulcers [cm], ulcerated surface, affected surface [%], and presence of narrowing) across 5 bowel segments (ie, rectum, descending and sigmoid colon, transverse colon, ascending colon, and ileum), where higher scores indicate more severe disease.
Percentage of Participants with Sustained Clinical and Endoscopic Remission at Week 54 | Week 54
  Sustained clinical and endoscopic remission is where a participant achieved clinical and endoscopic remission based on PCDAI and SES-CD scores at Weeks 14 and 54. Clinical remission is defined by PCDAI score ≤10. Endoscopic remission is defined as ≤4 with at least a 2-point reduction from Baseline and no sub-score >1 by SES-CD. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score ranges from 0 to 100, with higher scores indicating more active disease. The SES-CD score ranges from 0 to 56 and is the sum of 4 variables, size of ulcers [cm], ulcerated surface, affected surface [%], and presence of narrowing) across 5 bowel segments (ie, rectum, descending and sigmoid colon, transverse colon, ascending colon, and ileum), where higher scores indicate more severe disease.
Percentage of Participants with Corticosteroid-free Remission at Week 54 Based on PCDAI Score | Week 54
  Corticosteroid-free clinical remission is where participants achieves corticosteroid-free clinical remission based on PCDAI at Week 54 and has been off corticosteroids at least 12 weeks prior to and at Week 54. Clinical remission is defined by PCDAI score ≤10. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score ranges from 0 to 100, with higher scores indicating more active disease.
Percentage of Participants with Sustained Endoscopic Remission Based on SES-CD Score | Week 14
  Sustained endoscopic remission is where participants achieves endoscopic remission based on SES-CD ≤4 with at least a 2-point reduction from Baseline and no sub-score >1. The SES-CD evaluates 4 endoscopic variables (Size of ulcers, Ulcerated surface, Affected surface and Presence of narrowing). The score for each endoscopic variable is sum of values obtained for each segment. The SES-CD total is the sum of the four endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Percentage of Participants with Sustained Endoscopic Remission Based on SES-CD Score | Week 54
  Sustained endoscopic remission is where participants achieves endoscopic remission based on SES-CD ≤4 with at least a 2-point reduction from Baseline and no sub-score >1. The SES-CD evaluates 4 endoscopic variables (Size of ulcers, Ulcerated surface, Affected surface and Presence of narrowing). The score for each endoscopic variable is sum of values obtained for each segment. The SES-CD total is the sum of the four endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Percentage of Participants with Sustained Clinical Remission at Week 14 Based on PCDAI Score | Week 14
  Sustained Clinical Remission is where participants will achieve clinical remission based on PCDAI at Weeks 14 and 54. Clinical remission is defined by PCDAI score ≤10. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Percentage of Participants with Sustained Clinical Remission at Week 54 Based on PCDAI Score | Week 54
  Sustained Clinical Remission is where participants will achieve clinical remission based on PCDAI at Weeks 14 and 54. Clinical remission is defined by PCDAI score ≤10. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Serum Trough Concentrations of Vedolizumab Over Time | Predose and postdose at multiple time points (up to 54 weeks)
Percentage of Participants With Positive Antivedolizumab Antibodies | Pre-dose (up to 54 weeks)
Percentage of Participants With Positive Neutralizing Antivedolizumab Antibody Titers | Pre-dose (up to 54 weeks)
Sustained Clinical Response at Week 14 Based on PCDAI Score | Week 14
  Sustained clinical response is where a participant achieve clinical response based on PCDAI score ≤30 and reduction of the PCDAI by ≥15 points from Baseline. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Sustained Clinical Response at Week 54 Based on PCDAI Score | Week 54
  Sustained clinical response is where a participant achieve clinical response based on PCDAI score ≤30 and reduction of the PCDAI by ≥15 points from Baseline. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Percentage of Participants with Clinical Remission at Weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54 | Weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54
  Clinical remission is defined by PCDAI score < 10. The PCDAI was specifically designed for use in children. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT (adjusted for age and sex), ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Percentage of Participants with Change in Baseline in Clinical Response at Weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54 | Baseline, weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54
  Clinical Response is where participants achieves clinical response if PCDAI ≤30 with reduction in the PCDAI of ≥15 points from Baseline. The PCDAI includes a child-specific item: the height velocity variable as well as three laboratory parameters: HCT, ESR, and albumin level. The PCDAI score will range from 0 to 100, with higher scores indicating more active disease.
Percentage of Participants with at Least One Adverse Event (AE), Serious Adverse Event (SAE), and AE of special interest (AESI) | From first dose of study drug before each dose on dosing days through the Week 72
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have causal relationship with this treatment. AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether it is considered related to drug. SAE is any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to congenital anomaly/birth defect and/or is important medical event. An AESI (serious or non-serious) is one of scientific and medical concern specific to compound or program, for which ongoing monitoring and rapid communication by investigator. AESIs include- opportunistic infection, such as progressive multifocal leukoencephalopathy (PML), liver injury, malignancies, infusion-related reactions, hypersensitivity.
Change from Baseline in Weight | Baseline up to Week 54
  Change from in Baseline in weight will be calculated as: Weight at each study visit (up to Week 54) - Weight at Baseline.
Change from Baseline in Linear Growth Z-score | Baseline up to Week 54
  Linear growth Z-score will be calculated as: Z-score = (observed value - median value of the reference population)/ standard deviation value of reference population.
Change from Baseline in Tanner Stages at Week 54 | Week 54
  Tanner Stage is used to define physical measurements of sexual development based on external primary and secondary sex characteristics. Female and male participants are evaluated for breast development and genital development respectively and both genders for pubic hair distribution based on a 5-stage scale ranging from Stage I (prepubertal/preadolescent characteristics) to Stage V (mature or adult characteristics).

CONTACTS AND LOCATIONS:
Locations (95):
- United States (22):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - University of California San Francisco, San Francisco, California
  - I.H.S Health LLC, Kissimmee, Florida
  - Childrens Center For Digestive Healthcare, Atlanta, Georgia
  - Advocate Children's Hospital Park Ridge, Park Ridge, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - MNGI Digestive Health, PA, Minneapolis, Minnesota
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Goryeb Children's Hospital, Morristown, New Jersey
  - The Steven and Alexandra Cohen Childrens Medical Center of New York - BRANY - PPDS, New Hyde Park, New York
  - University of Rochester Medical Center PPDS, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Texas Children's Hospital, Houston, Texas
  - Carilion Children's Tanglewood Center, Roanoke, Virginia
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Brussel - PIN, Jette, Brussels Capital
  - UZ Leuven, Leuven, Vlaams Brabant
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- China (4):
  - Beijing Children Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Henan Children's Hospital(Zhengzhou Children's Hospital), Zhengzhou, Henan
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Children's Hospital Zhejiang UniversitySchool of Medicine, Hangzhou, Zhejiang
- Croatia (3):
  - Klinika Za Djecje Bolesti Zagreb, Zagreb, City of Zagreb
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - University Hospital Centre Split, Split
- Czechia (3):
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha, Hlavni Mesto
  - Fakultni Thomayerova Nemocnice, Prague, Praha, Hlavni Mesto
  - Fakultni nemocnice Ostrava, Ostrava
- Greece (3):
  - Attikon University General Hospital, Athens, Attica
  - Children's Hospital "Agia Sofia", Athens
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Semmelweis Egyetem, Budapest
- Israel (7):
  - Schneider Childrens Medical Center of Israel Petah Tikvah PIN, Petah Tikva, Central District
  - Tel Aviv Sourasky Medical Center PPDS, Jerusalem, Jerusalem
  - Soroka University Medical Centre, Beersheba
  - Rambam Medical Center - PPDS, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem
- Italy (6):
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda USL di Bologna, Bologna, Emilia-Romagna
  - Sapienza University of Rome, Rome, Lazio
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - Universita degli Studi di Padova, Padua, Veneto
- Japan (4):
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - National Center for Child Health and Development, Setagaya-Ku, Tokyo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Kaunas County
  - Vilnius University Hospital Santaros Klinikos, Vilnius, Vilnius County
- Poland (10):
  - Uniwersytecki Szpital Dzieciecy, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Masovian Voivodeship
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Gornoslaskie Centrum Zdrowia Dziecka Im. Sw. Jana Pawla II Spsk Nr 6 Sum W Katowicach, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Slovakia (2):
  - Detska fakultna nemocnica s poliklinikou Banska Bystrica, Banská Bystrica
  - Narodny ustav detskych chorob, Bratislava
- South Korea (4):
  - Kyungpook National University Chilgok hospital, Daegu, Daegu Gwang'yeogsi
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Seoul National University Hospital, Seongnam
  - Samsung Medical Center - PPDS, Seoul
- Spain (5):
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat, Barcelona
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Infantil Universitario Nino Jesus - PIN, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Materno Infantil, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (6):
  - Kings College Hospital, London, London, City of
  - Great Ormond Street Hospital (GOSH), London, London, City of
  - Noahs Ark Childrens Hospital for Wales - PPDS - PIN, Cardiff, South Glamorgan
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Barts Health NHS Trust, London
  - Royal Manchester Children's Hospital - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/60423b8eeb9d7e001f5bc61f